CLINICAL TRIAL: NCT02850991
Title: A Multicenter, Prospective, Randomized, Phase III Trial Evaluating High-dose Versus Standard-dose Radiation With Concurrent Chemotherapy for Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Different Radiation Dose With Concurrent Chemotherapy for Thoracic Esophageal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Anhui Shi, MD, MD, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESR-15-11224
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer, radiation, chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: High dose radiation plus chemotherapy of paclitaxel and carboplatin vs standard dose radiation plus chemotherapy of paclitaxel and carboplatin.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-dose (Experimental): concurrent chemoradiotherapy High-dose RT:59.4 Gy in 33 fractions, 1.8 Gy per fraction, 5days/week; CT: Paclitaxel 50 mg/m2 D1+carboplatin AUC (area under curve) =2 D1, weekly for 6 weeks.
  After that, patients receive consolidative platinum-based 3-week chemotherapy for 2 cycles.
  Interventions: Radiation: High-dose
- Standard-dose (Active Comparator): concurrent chemoradiotherapy Standard-dose RT:50.4 Gy in 28 fractions, 1.8Gy per fraction, 5days/week; CT: Paclitaxel 50 mg/m2 D1+carboplatin AUC (area under curve) =2 D1, weekly for 6 weeks.
  After that, patients receive consolidative platinum-based 3-week chemotherapy for 2 cycles.
  Interventions: Radiation: Standard-dose

INTERVENTIONS:
Radiation: High-dose — Drug: concurrent chemotherapy with radiation paclitaxel plus carboplatin are used weekly in both arms
  Arms: High-dose
Radiation: Standard-dose — Drug: concurrent chemotherapy with radiation paclitaxel plus carboplatin are used weekly in both arms
  Arms: Standard-dose

SUMMARY:
Definitive chemoradiation is the standard treatment for locally advanced esophageal cancer. NCCN (National Comprehensive Cancer Network) recommends radiation dose of 50-50.4 Gy as the definitive radiation dose for esophageal cancer with definitive chemo-radiation. However, as many studies in China showed that the most common recurrence site after definitive chemo-radiation was within the radiation region. But there have not been large randomized clinical trials to investigate the optimal radiation dose with concurrent chemotherapy for esophageal cancer in China. The purpose of this clinical trial is to investigate the optimal radiation dose for thoracic esophageal squamous cell cancer with definitive concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if high-dose radiation with concurrent chemotherapy increases overall survival for thoracic esophageal squamous cell carcinoma

SECONDARY OBJECTIVES:

I. To evaluate if high-dose radiation with concurrent chemotherapy increased progression-free survival for thoracic esophageal squamous cell carcinoma II.To evaluate if high-dose radiation with concurrent chemotherapy increased local control for thoracic esophageal squamous cell carcinoma

OUTLINE:

Patients are randomized to one of the two treatment arms

ARM 1:Patients receive high-dose radiation with concurrent chemotherapy.High-dose RT:59.4 Gy in 33 fractions, 1.8 Gy per fraction, 5days/week.concurrent chemotherapy: Paclitaxel 50mg/m2 D1+carboplatin AUC (area under curve) =2 D1, weekly for 6 weeks. After that, patients receive consolidative platinum-based 3-week chemotherapy for 2 cycles.

ARM 2:Patients receive standard-dose radiation with concurrent chemotherapy.Standard-dose RT:59.4 Gy in 33 fractions, 1.8 Gy per fraction, 5days/week . Concurrent chemotherapy: Paclitaxel 50 mg/m2 D1+carboplatin AUC (area under curve) =2 D1, weekly for 6 weeks. After that, patients receive consolidative platinum-based 3-week chemotherapy for 2 cycles.

After completion of study therapy, patients are followed up every 3-4 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Age: 18-75 years
3. Histological or cytologic diagnosis of esophageal squamous cell carcinoma within one month. Clinical stage T1-4 N0-1 M0-1a (AJCC 6th edition）. Supraclavicular lymphatic metastasis or abdominal lymph node metastasis for mid-thoracic also can be included
4. Karnofsky performance status scores: ≥70
5. Without any prior anticancer therapy
6. BMI≥18kg/m2 or weight loss ≤5% within 3 months
7. Adequate marrow function (within 7 days): White blood cell ≥ 3×109/L,Neutrophils (ANC) ≥1.5×109/L, Platelet count ≥100×109/L, Hemoglobin ≥90g/L. Normal hepatic and renal function (within 14 days): Total bilirubin <1.5 x upper limit of normal (ULN), Alanine aminopeptidase and Aspartase aminotransferase ≤ 2.5 x ULN, creatinine ≤ 1.5xULN
8. Normal cardiac and pulmonary function: Forced expiratory volume at one second (FEV1) ≥1.0 L or FEV1/FVC ≥ 50% pre FEV1; No myocardial infarction within 1 year; no symptomatic heart disease, including myocardial ischemia, congestive heart failure or uncontrolled arrhythmias, roughly normal electrocardiogram; LVEF ≥ 50%，or can receive chemoradiotherapy assessed by cardiologists

Exclusion Criteria:

1. Other or mixed pathological type
2. The second primary tumor of esophageal cancer located outside the radiation area
3. Biopsy-proven invasion of the tracheobronchial tree or tracheoesophageal fistula
4. Mid-thoracic esophageal cancer with supraclavicular lymphatic metastasis and abdominal lymph node metastasis; other metastasis
5. Within 2cm of the gastroesophageal junction
6. Prior chemotherapy, prior thoracic radiation, surgical resection or target therapy of the primary tumor
7. Significant medical or psychiatric illnesses that in the physician's judgment (uncontrolled coronary heart disease, cardiomyopathy and/or heart failure requiring hospitalization. Uncontrolled hypertension or history of myocardial infarction within one year. Uncontrolled diabetes mellitus. Acute bacterial or fungal infection requiring intravenous antibiotics. Acute exacerbation of chronic obstructive pulmonary disease (COPD) or other pulmonary disease requiring hospitalization influencing tumor treatment
8. Refused to sign informed consent form
9. Concurrent pregnancy or lactation
10. History of a second malignancy other than nonmelanoma skin cancer, and cervical cancer in situ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-04; Primary Completion 2019-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 5 years

SECONDARY OUTCOMES:
Progression-free survival | 5 years

OTHER OUTCOMES:
local control rate, recurrence pattern | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anhui Shi, MD., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided